CLINICAL TRIAL: NCT05757401
Title: Sleep Quality After Cesarean Delivery Under Spinal Anesthesia With Intrathecal Morphine and Related Factors
Brief Title: Sleep Quality After Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 831/2565(IRB1); Si 898/2022 (Registry Identifier: Siriraj Institutional Review Board)
Record Dates: First submitted 2023-01-26; First posted 2023-03-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Section Complications; Sleep Disturbance; Perioperative Complication
Keywords: cesarean delivery; sleep quality; Perioperative complication
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgery causes poor sleep quality for several reasons eg. increasing stress hormonal production, pain, starvation, and environmental procedure namely noise, light, and nursing procedures. Poor sleep quality also brings numerous side effects including delirium, delayed recovery, and affect breastfeeding. We, therefore, aim to elucidate the incidence of poor sleep quality in parturients undergoing cesarean delivery in the early postoperative period and investigate the factors involving poor sleep conditions.

DETAILED DESCRIPTION:
Surgery causes poor sleep quality for several reasons eg. increasing stress hormonal production, pain, starvation, and environmental procedure namely noise, light, and nursing procedures. Postoperative pain after cesarean delivery can be found as high as 70 percent in the first postoperative pain. Also, the side effect of anesthetic may cause poor sleep quality such as itching, nausea, and vomiting.

Poor sleep quality brings numerous side effects including delirium, delayed recovery, and affect breastfeeding. The data on obstetric patients sleep quality in the early postoperative period is scarce. We, therefore, aim to elucidate the incidence of poor sleep quality in parturients undergoing cesarean delivery in the early postoperative period and investigate the factors involving poor sleep conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age >,= 18 years, undergoing cesarean delivery
* Receive spinal anesthesia with local anesthetic drug and intrathecal morphine
* Understand Thai

Exclusion Criteria:

* Patients receive epidural block or nerve block
* Patients require conversion to general anesthesia with any reasons
* Patients require endotracheal intubation with any reasons
* Patients admit to intensive care unit in postoperative period
* Patients with the end of operation at the time 24.00-6.00 AM

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parturients age >,= 18 years old undergoing cesarean delivery
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Sleep quality | 24 hours postoperative
  Sleep quality at the first postoperative day evaluated by Richard Campbell Sleep Questionaire- Thai version

SECONDARY OUTCOMES:
Nausea and vomiting score | 24 hours postoperative
  Nausea and vomiting score; 0 = no symptom, 1= mild symptom nausea and no vomiting, 2 = vomiting 1-2 times, 3 = severe vomiting or needed treatment
Itching | 24 hours postoperative
  Itching score; 0 = no itching, 1= mild itching, 2 = severe itching or needed treatment
Postoperative pain | 24 hours postoperative
  11-point Numerical rating score (NRS) pain scale ranging from 0-10, 0= no pain, 10 = severe pain
EQ-5D-5L | 24 hours postoperative
  Quality of life evaluated by EuroQol group-5 Dimentions-5 levels questionnaire (EQ-5D-5L)- Thai version
LATCH score | 24 hours postoperative and at the discharge day
  LATCH score comprise of 5 components: Latch, Audible swallowing, Type of nipple, Comfort and Hold- each component scored from 0-2, A total of less than 8 is considered unsatisfactory
Length of hospital stay | Through the study completion an average 3-5 days
  Length of hospital stay
Neonatal weight | Postoperative day 1 and day 3
  The weight of neonate

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Anesthesiology department, Siriraj hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
The data-sharing plan is undecided.

REFERENCES:
- [Result] Jintadawong T, Nivatpumin P, Swaengrujitham M, Punchuklang W, Lertbunnaphong T. Sleep quality after caesarean delivery: associated factors and effects on quality of life and early breastfeeding. Ann Med. 2025 Dec;57(1):2582917. doi: 10.1080/07853890.2025.2582917. Epub 2025 Nov 12. PMID 41229134